CLINICAL TRIAL: NCT00646009
Title: A Randomized, Multicenter, Placebo and Active-controlled, Single-dose, 4-period, Crossover Study to Evaluate the Bronchodilating Effect of SYMBICORT pMDI Versus Advair Diskus and Ventolin HFA.
Brief Title: Symbicort Onset of Action 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SD-039-0733; D5896C00733
Record Dates: First submitted 2008-03-26; First posted 2008-03-28 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Asthma
Keywords: asthma; adults; Symbicort; budesonide/formoterol; Advair Diskus; Ventolin
MeSH Terms: conditions — Asthma | interventions — Budesonide, Formoterol Fumarate Drug Combination; Fluticasone-Salmeterol Drug Combination; Albuterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): budesonide/formoterol
  Interventions: Drug: budesonide/formoterol
- 2 (Active Comparator): fluticasone/salmeterol
  Interventions: Drug: fluticasone/salmeterol
- 3 (Active Comparator): albuterol
  Interventions: Drug: albuterol

INTERVENTIONS:
Drug: budesonide/formoterol
  Other Names: Symbicort
  Arms: 1
Drug: fluticasone/salmeterol
  Other Names: Advair Diskus
  Arms: 2
Drug: albuterol
  Other Names: Ventolin
  Arms: 3

SUMMARY:
The purpose of this study is to compare the early onset of effect of Symbicort compared to Advair Diskus and Ventolin in adults with asthma

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Diagnosis of asthma and baseline lung function test results as determined by the protocol
* Required and received inhaled corticosteroids within timeframe and doses specified in the protocol

Exclusion Criteria:

* Severe asthma or asthma that is markedly effected by seasonal factors
* Has required and received non-inhaled corticosteroids within the previous 4 weeks, has sensitivity to drugs specified in the protocol or requires treatment with beta-blockers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2003-03; Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
FEV1 3 minutes post dose | 4 assessments across 4 visits whilst on treatment (visits may be between 3 and 14 days apart)

SECONDARY OUTCOMES:
12 hour serial FEV1 | 4 assessments across 4 visits whilst on treatment (visits may be between 3 and 14 days apart)
Patients perception of effect | Patients perception of effect

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Bonuccelli, Study Director — AstraZeneca